CLINICAL TRIAL: NCT04456023
Title: A Phase II, Single-arm, Multicenter Trial to Evaluate the Efficacy and Safety of Tisagenlecleucel in Chinese Adult Patients With Relapsed or Refractory Diffuse Large B-cell Non-Hodgkin Lymphoma (DLBCL)
Brief Title: Study of Tisagenlecleucel in Chinese Adult Patients With Relapsed or Refractory Diffuse Large B-cell Non-Hodgkin Lymphoma (DLBCL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was cancelled before enrolling any patients for business related reasons.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019C2203
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: Diffuse Large B-cell Lymphoma; double/triple hit lymphoma; relapsed/refractory; tisagenlecleucel; CTL019; Chinese
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): All patients eligible for treatment with tisagenlecleucel will receive a single dose of tisagenlecleucel.
  Interventions: Biological: Tisagenlecleucel

INTERVENTIONS:
Biological: Tisagenlecleucel — A single intravenous (i.v.) infusion of 0.6 - 6.0×10^8 CAR positive viable T cells.
  Other Names: CTL019

SUMMARY:
This is a multi-center, phase II study to evaluate the efficacy and safety of CTL019 in Chinese adult patients with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
Disease assessments will be performed at screening, after bridging, 1, 3, 6, 9 and 12 months after tisagenlecleucel infusion, and every 6 months in the second year, and annually up to 60 months after infusion. Efficacy will be assessed until progression; safety will be assessed throughout the study. A long term follow-up up to 15 years after CTL019 infusion will continue under a separate protocol (CCTL019A2205B)(NCT02445222).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Patients must be ≥18 years of age at the time of ICF signature
3. Histologically confirmed DLBCL at last relapse (including DLBCL transformed from follicular lymphoma and double-triple hit lymphoma)
4. Relapsed or refractory disease after at least 2 lines of systemic therapy, including anti-CD20 antibody and an anthracycline, or having failed or being ineligible for autologous HSCT
5. ECOG performance status that is either 0 or 1 at screening
6. Measurable disease at time of enrollment:

   * Nodal lesions greater than 15 mm in the long axis, regardless of the length of the short axis or
   * Extra nodal lesion (outside lymph node or nodal mass, but including liver and spleen) at least 10 mm in long and short axis
7. Adequate organ function
8. Must have a leukapheresis material of non-mobilized cells available for manufacturing

Exclusion Criteria:

1. Prior treatment with anti-CD19 therapy, adoptive T cell therapy, or any prior gene therapy product
2. Primary mediastinal large B-cell lymphoma, EBV+ DLBCL, Richter's transformation, Burkitt lymphoma, primary DLBCL of CNS, T cell / histiocyte rich large B-cell lymphoma, primary cutaneous DLBCL.
3. Eligible for and consenting to autologous HSCT
4. Prior allogeneic SCT
5. Active CNS involvement by disease under study, except if the CNS involvement has been effectively treated (i.e. patient is asymptomatic) and local treatment was greater than 4 weeks before enrollment
6. Active neurological autoimmune or inflammatory disorders (e.g. Guillain-Barre syndrome)
7. Investigational medicinal product within the last 30 days or five half-lives (whichever is longer) prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Complete Response (CR) and Partial Response (PR) according to the Lugano classification as determined by the Investigator.

SECONDARY OUTCOMES:
Duration of Response (DOR) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Time from CR or PR, whichever occurs first, to relapse or death due to DLBCL.
Time to response (TTR) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Time from tisagenlecleucel infusion to CR or PR, whichever occurs first.
Progression-Free Survival (PFS) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Time from tisagenlecleucel infusion to the first documented disease progression or death due to any cause.
Event free survival (EFS) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Time from tisagenlecleucel infusion to the first documented disease progression or relapse, new treatment for lymphoma or death due to any cause.
Overall Survival (OS) | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Time from tisagenlecleucel infusion to death due to any cause.
Number of Participants with On-Treatments Adverse Events, Serious Adverse Events, and Deaths | From first dosing (single administration, Day 1) up to End of Study Visit (EOS), an average of 60 Months
  Analysis of absolute and relative frequencies for treatment emergent AE, SAE and Deaths by primary System Organ Class (SOC) through the monitoring of relevant clinical and laboratory safety parameters.
Tisagenlecleucel immunogenicity (humoral) | Up to Month 60
  The humoral immunogenicity assay will be evaluated to measure the antibody titers specific to the tisagenlecleucel molecule prior to and following infusion.
Tisagenlecleucel immunogenicity (cellular) | Up to Month 60
  The cellular immunogenicity assay will be evaluated to assess the presence of T lymphocytes activated by the tisagenlecleucel protein.
In vivo cellular PK profile of tisagenelecleucel | Up to Month 60
  qPCR and flow cytometry to measure tisagenlecleucel transgene concentration in blood, bone marrow and other matrices/tissues.
Concentration of Tocilizumab PK in tocilizumab treated subjects during CRS | Up to Day 7 after tocilizumab infusion
  Concentration of Tocilizumab
Serum cytokines (IL-10, interferon gamma, IL-6, CRP and ferritin) | Up to Month 60
  Concentration of soluble factors (IL-10, interferon gamma, IL-6, CRP and ferritin) will be listed and summarized by participant and time point.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338